CLINICAL TRIAL: NCT02545231
Title: Effect of Low-dose vs. High-dose Pitavastatin on In-stent Restenosis, Endothelial Function, Circulating microRNAs, and Cardiovascular Events in Patients With Coronary Artery Disease Requiring Stent Implantation: OCT and NIRS Comparison
Brief Title: Effect of Low-dose vs. High-dose Pitavastatin on In-stent Restenosis
Acronym: ELEVATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pitavastatin
Record Dates: First submitted 2015-09-02; First posted 2015-09-09 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Atherosclerosis; Neointima; Angina
MeSH Terms: conditions — Atherosclerosis; Neointima; Angina Pectoris | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose 1mg pitavastatin (Active Comparator): pitavastatin 1mg which is considered low dose statin will be administered for 36 months
  Interventions: Drug: Pitavastatin 1mg; Drug: Placebo
- High dose 4mg pitavastatin (Active Comparator): pitavastatin 4mg which is considered high dose statin will be administered for 36 months
  Interventions: Drug: Pitavastatin 4mg; Drug: Placebo

INTERVENTIONS:
Drug: Pitavastatin 1mg — To compare different doses of statins on atherosclerosis progression and neointimal hyperplasia
  Other Names: Livalo 1mg
  Arms: Low dose 1mg pitavastatin
Drug: Pitavastatin 4mg — To compare different doses of statins on atherosclerosis progression and neointimal hyperplasia
  Other Names: Livalo 4mg
  Arms: High dose 4mg pitavastatin
Drug: Placebo — To compare different doses of statins on atherosclerosis progression and neointimal hyperplasia

SUMMARY:
To compare low dose (1mg) pitavastatin and high dose (4mg) pitavastatin on neointimal hyperplasia and atherosclerosis progression by using optical coherence tomography (OCT) and near-infrared spectroscopy (NIRS) at 12 months follow-up and on clinical adverse cardiovascular events during 3-year follow-up.

DETAILED DESCRIPTION:
* Patients with non-ST elevation ACS will be randomized into pitavastatin 1mg or 4mg after everolimus-eluting stent implantation with OCT and NIRS study.
* 12 months follow-up coronary angiography with OCT and NIRS will be performed to compare neointimal hyperplasia and atherosclerosis progression.
* 36 months clinical follow-up for major adverse cardiovascular events (cardiac death, all-cause death, myocardial infarction, stroke, target lesion revascularization) will be compared.
* Safety issues such as bleeding rates, abnormal liver function will be compared

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Patients between the age of 30 to 79
3. Non-ST elevation Acute coronary syndrome with successful everolimus eluting stent implantation (with TIMI flow grade 3 after the procedure)

Exclusion Criteria:

1. Hypersensitivity to pitavastatin
2. Unable to perform OCT and NIRS
3. Serum creatinine > 2.0 mg/dL.
4. Steroid or hormone replacement therapy
5. Hemoglobin A1c >9%
6. Type 1 diabetes
7. Decreased serum platelet level (< 100,000/uL)
8. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin
9. Life expectancy less than a year
10. Renal failure requiring dialysis or anticipated need for dialysis during the course of the study
11. Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study
12. Involvement in the planning and/or conduct of the study
13. Left ventricular ejection fraction < 40%
14. Hepatic dysfunction (aspartate aminotransferase or alanine aminotransferase > twice the upper limit)
15. Gastrointestinal disorder such as Crohn's disease
16. Alcohol abuse
17. Known pregnancy, breast-feeding, or intend to become pregnant during the study period

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2013-02; Primary Completion 2018-12 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Neointimal volume with OCT (mm3 per 1mm) and lipid volume with NIRS (the maximal lipid core burden index (LCBI) in 4 mm segment during 12 months of treatment | 12 months for OCT and NIRS
  OCT will measure neointimal volume in every mm interval and will be averaged by dividing the total neointimal volume with the number of the segment analyzed. LCBI is the lipid volume index which is calculated automatically by the device, and LCBI > 400 is considered high lipid volume.

SECONDARY OUTCOMES:
Rates of major adverse cardiovascular events during 12 months follow-up | 12 months for clinical events
  Major adverse cardiovascular events include all-cause death, cardiovascular death, myocardial infarction, stroke, target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Do-Sun Lim, MD, PhD, Study Chair — Korea University Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jeong HS, Hong SJ, Son S, An H, Kook H, Joo HJ, Park JH, Yu CW, Lim DS. Incidence of new-onset diabetes with 1 mg versus 4 mg pitavastatin in patients at high risk of developing diabetes during a 3-year follow-up. Cardiovasc Diabetol. 2019 Nov 21;18(1):162. doi: 10.1186/s12933-019-0969-z. PMID 31752850
- [Derived] Lim JW, Jeong HS, Hong SJ, Kim HJ, Kim YC, Kang BG, Jeon SM, Cho JY, Lee SH, Joo HJ, Park JH, Yu CW. Effects of lowest-dose vs. highest-dose pitavastatin on coronary neointimal hyperplasia at 12-month follow-up in type 2 diabetic patients with non-ST elevation acute coronary syndrome: an optical coherence tomography analysis. Heart Vessels. 2019 Jan;34(1):62-73. doi: 10.1007/s00380-018-1227-0. Epub 2018 Jul 25. PMID 30047013